CLINICAL TRIAL: NCT00844441
Title: Pilot Study of Feasibility, Safety, and Economics of Early Discharge and Outpatient Management of Adult Patients Following Intensive Induction Chemotherapy for Myelodysplastic Syndrome and Non-APL Acute Myeloid Leukemia
Brief Title: Early Discharge and Outpatient Care After Chemotherapy in Patients With Myelodysplastic Syndrome or Acute Myeloid Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Roland Walter, Fred Hutchinson Cancer Research Center
Purpose: Health Services Research
Other Study IDs: 2300.00; P30CA015704 (NIH); FHCRC-2300.00; IR 6845; CDR0000631997 (Registry Identifier: PDQ)
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute eosinophilic leukemia; adult acute monocytic leukemia (M5b); adult acute megakaryoblastic leukemia (M7); adult acute basophilic leukemia; acute myeloid leukemia with multilineage dysplasia following myelodysplastic syndrome; adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b)
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Basophilic, Acute; Leukemia, Erythroblastic, Acute

INTERVENTIONS:
Other: medical chart review
Other: questionnaire administration
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Gathering information about patients with myelodysplastic syndrome or acute myeloid leukemia who are discharged after finishing chemotherapy, or who stay in the hospital until blood counts return to normal, may help doctors learn more about a patient's quality of life, use of medical services, and the cost of these services.

PURPOSE: This clinical trial is studying early discharge and outpatient care in patients who have undergone chemotherapy for myelodysplastic syndrome or acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the death rate in patients with myelodysplastic syndromes or acute myeloid leukemia who are discharged after completion of induction chemotherapy vs those who remain in the hospital until blood counts recover.

Secondary

* To determine the proportion of patients who meet the early discharge criteria after completion of induction chemotherapy.
* To compare the costs incurred by patients who are discharged early vs those who are discharged only after blood counts recover.
* To compare resource utilization (e.g., transfusions) among these patients.
* To compare the quality of life of these patients.

OUTLINE: Within 72 hours after completion of induction chemotherapy, patients are either discharged from the hospital or remain in the hospital until their blood counts recover.

Patients receive standard supportive care after completion of induction chemotherapy either in the hospital or as an outpatient. Outpatients are seen by a registered nurse or physician assistant ≥ 3 times weekly and by a physician at least once weekly.

A medical chart review is conducted to obtain information about medical complications (e.g., neutropenic fever, documented infections, bleeding, reasons for hospitalization) and use of medical resources. Patients complete the MDA Symptom Inventory and the EORTC QLQ-C30 questionnaire periodically to assess quality of life. Costs associated with inpatient and outpatient care are evaluated using electronic billing information from the University of Washington Medical Center and Seattle Cancer Care Alliance.

After completion of the study, patients are followed up for 1 month.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following:

  * Myelodysplastic syndromes
  * Acute myeloid leukemia (AML)

    * No acute promyelocytic leukemia with t(15;17)(q22;q12), PML/RAR, or other variants
* Planning to undergo AML-like intensive induction chemotherapy (e.g., "7+3" or regimen with similar or higher intensity) for untreated or relapsed disease within 1 week after study entry OR has started therapy within the past 72 hours

PATIENT CHARACTERISTICS:

* No hypersensitivity or allergy to fluoroquinolones, triazoles, or acyclovir
* ECOG/WHO/ZUBROD performance status 0-1*
* Total bilirubin ≤ 2.5 times upper limit of normal (ULN) (unless elevation is thought to be due to Gilbert's syndrome or hemolysis)*
* AST and ALT ≤ 1.5 times ULN*
* Serum creatinine ≤ 1.5 times ULN*
* No clinical evidence of congestive heart failure*
* No active bleeding*
* Not refractory to platelet transfusions (e.g., due to HLA-alloimmunization)*
* No requirement for IV antimicrobial therapy*
* Agrees to undergo close follow-up that includes ≥ 3 visits per week at the Seattle Cancer Care Alliance (SCCA)*
* Has a confirmed reliable caregiver and transportation*
* Confirmed temporary or permanent residency within a 30-minute commute from the University of Washington (UW) Medical Center/SCCA*
* Has identified a UW/SCCA hematologist/oncologist who is willing to care for the patient in the outpatient clinic* NOTE: *Additional criteria for early discharge from the hospital

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-09 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Death rate in patients discharged after completion of induction chemotherapy
Rate of successful discharge of patients who meet medical discharge criteria
Costs associated with outpatient vs inpatient treatment
Medical resources used with outpatient vs inpatient treatment

CONTACTS AND LOCATIONS:
Overall Officials: Roland Walter, MD, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (3):
- United States (2):
  - Oregon Health and Science University, Portland, Oregon
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Clinical Cancer Research Center at University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Walter RB, Lee SJ, Gardner KM, Chai X, Shannon-Dorcy K, Appelbaum FR, Estey EH. Outpatient management following intensive induction chemotherapy for myelodysplastic syndromes and acute myeloid leukemia: a pilot study. Haematologica. 2011 Jun;96(6):914-7. doi: 10.3324/haematol.2011.040220. Epub 2011 Mar 10. PMID 21393334